CLINICAL TRIAL: NCT05062785
Title: Phase 1, Open Label Dose-Finding Study of Intranasal Insulin in Healthy Participants
Brief Title: Dose-Finding Study of Intranasal Insulin in Healthy Participants Insulin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Silbergleit (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Robert Silbergleit, Professor of Emergency Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HUM00171279
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Healthy
Keywords: Healthy participants; intranasal insulin
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: For every 6 participants, iterations of a Bayesian model will be performed to associate the administered dose with the frequency of dose-limiting hypoglycemia or other adverse events. The model will adaptively reallocate the dose increments for the next 6 participants. To provide more precise and reproducible estimates of dose-limiting toxicity, the trial will modify the size of dose increments based on the developing model to allocate more administrations to areas of the model with greatest uncertainty, or to higher doses in the absence of dose-limiting hypoglycemia.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal insulin (Experimental): A total of 11 possible doses will be tested, ranging from 0 to 1000 U insulin.
  Interventions: Drug: Intranasal insulin

INTERVENTIONS:
Drug: Intranasal insulin — This will be given intranasally at differing doses depending on study day. A total of 11 possible doses will be tested, ranging from 0 to 1000 U insulin. Each volunteer will come for 5 visits.
  On the first treatment day participants will receive placebo (sterile water) in each nostril followed by a 4-hour observation period. After this observation period participants will receive the initial dose of insulin squirted in each nostril followed by a a 4 hour observation period. Participants will have at least 7 days in between the other 4 visits. Subsequent visits will include increased doses of insulin (depending on how this is tolerated) and will take approximately 4 hours at these visits.
  Other Names: HUMULIN R U-500

SUMMARY:
This study is to determine the safety and tolerability of regular insulin (Humulin R) when given intranasally (as drops in nostrils).

Healthy participants will be enrolled to determine the maximum tolerated dose of intranasal insulin.

DETAILED DESCRIPTION:
This is being studied because intranasal insulin may be a way to prevent the brain injury that occurs after a cardiac arrest. Cardiac arrest is a life-threatening condition in which the heart suddenly stops beating and there is no blood flow to the body. If cardiac arrest is not treated immediately, it causes sudden death. Even when immediate treatment gets the heart beating again, many victims remain comatose and die later from brain injury. Nasal insulin, given immediately after a cardiac arrest may prevent or reduce brain injury. Nasal insulin reduces brain injury in animal experiments, and has been used to try to improve brain degeneration in patients with Alzheimer's disease. However, cardiac arrest patients may need higher doses than patients with Alzheimer's disease, therefore, this study is to examine those higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Good health based on medical history, physical exam, and routine laboratory testing.
* Female participants must have negative urine pregnancy test or be surgically sterilized or postmenopausal. Criteria for menopause are surgical menopause (hysterectomy, oophorectomy) or age > 45 years with the absence of menses for greater than 12 months. Tubal ligation with menses within the past 12 months is not considered to be surgical sterilization.
* Body mass index (BMI) between 18 kilogram / square meter (kg/m2) and 35 kg/m2.
* Willing and able to stay at the clinical research facility as required by the protocol
* Willing and able to comply with the investigational nature of the study and able to communicate well with investigators
* Ability to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines

Exclusion Criteria:

* Known allergy to insulin.
* Preexisting diabetes.
* Current or previous use of diabetes medication or insulin.
* Any nasal disease or congestion that may interfere with intranasal drug absorption.
* Baseline hypoglycemia (blood glucose ≤ 65 mg/dL) or hyperglycemia (blood glucose > 200 mg/dL) as evident from the screening labs.
* Active serious disease, such as liver disease, kidney disease, uncontrolled hypertension, clinically significant hypokalemia, and significant or unstable medical illness
* Blood donation in excess of 500 milliliter (mL) within 60 days prior to the first dose of study medication.
* Treated with an investigational drug within 30 days.
* Individuals with inadequate venous access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Severe Hypoglycemia as defined by blood glucose < 45 milligrams per deciliter (mg/dL) | Up to 4 hours after drug administration
  Severe Hypoglycemia will be considered a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Change in blood glucose | Baseline, up to 4 hours after drug administration
Change in serum insulin | Baseline, up to 4 hours after drug administration
Change in serum C-peptide levels | Baseline, up to 4 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Robert Silbergleit, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No